CLINICAL TRIAL: NCT03892057
Title: Internet-based Positive Psychological Intervention for Hispanic/Latino Adult With Hypertension in a Primary Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Rosenfeld Heart Foundation Grant (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08776
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Uncontrolled Hypertension; Cardiovascular Risk Factor
Keywords: Hispanics/Latinos; Underserved Population; Internet-based

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blind to intervention assignment and will only collect clinical data at baseline, 5-, and 12-weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based Positive Psychological Intervention (Experimental): The investigator's culturally-tailored internet-based Positive Psychology (PP) Intervention is a non-pharmacotherapy approach aimed at increasing positive emotional experiences by teaching individuals to engage in intentional activities known to increase psychological and emotional well-being through targeting of constructs such as optimism, gratitude, mindfulness/relaxation, and resilience.
  Interventions: Behavioral: Internet-based Positive Psychological Intervention
- Attention Control Group (No Intervention): Participants will complete computerized surveys to document the frequency of positive and negative emotions experienced in daily life. The attention control group will be given the option to access our positive psychological intervention and associated content via the web at the conclusion of the 12-week data collection phase.

INTERVENTIONS:
Behavioral: Internet-based Positive Psychological Intervention — The investigator's culturally-tailored internet-based Positive Psychology Intervention is a non-pharmacotherapy approach aimed at increasing positive emotional experiences by teaching individuals to engage in intentional activities known to increase psychological and emotional well- being, e.g., mindfulness/meditation. The current 5-week Internet-based intervention will be delivered via a secure website which participants will access at home (or in a public setting with Wi-Fi) using an assigned username and password. The on-line program includes didactic material and "home practice" with participants logging into the website 3-4 times per week for 15 to 20 minute sessions. In addition to weekly on-line instruction, participants are assigned homework as a means of incorporating skills learned into their day-to-day activities.
  Other Names: Positive Affect Intervention
  Arms: Internet-based Positive Psychological Intervention

SUMMARY:
The largest epidemiologic study of Hispanic/Latino participants thus far, i.e., the Hispanic Community Health Study/Study of Latinos (HCHS/SOL) documented that 80% of men and 71% of women have at least one major cardiovascular disease (CVD) risk factor. The American Heart Association emphasizes that current CVD prevention efforts are sparse and ineffectual in minority populations and acknowledges the need for new and more effective disease prevention strategies. This proof-of-concept study and pilot randomized clinical trial seeks to implement and evaluate a novel internet-based 5-week Positive Psychology (PP) Intervention (compared to an attention control condition) in Hispanic/Latino adults with uncontrolled hypertension, i.e., elevated 24-hour ambulatory blood pressure, with primary interest in testing efficacy for clinically meaningful improvements in cardiovascular function.

DETAILED DESCRIPTION:
The study features piloting of a randomized trial to determine whether an internet-based positive psychology (PP) intervention is associated with greater improvements in blood pressure compared to an attention control condition. The pilot trial additionally evaluates the efficacy of the internet-based PP intervention with respect to psychological well-being, hypertension-related health behaviors, autonomic cardiac control, and high-sensitivity C-reactive protein. Serum blood assays will facilitate exploration of mechanistic indicators linking psychological well-being to cardiac functioning.

ELIGIBILITY:
Inclusion Criteria:

* Hispanics/Latinos recruited from UI Health Pilsen Family Health Center Lower West
* Aged ≥18
* Fluent in English or Spanish with ≥8th grade education
* Elevated sitting blood pressure (≥140/90)
* Ability to read and understand the informed consent
* Ability to access internet from home or in public setting (note, tablet PCs will be made available to all enrolled participants at no charge), and
* Self-reported comfort in with handling of a table computer and website navigation.

Exclusion Criteria:

* Cognitive impairment denoting dementia (assessed using the Short Portable Status Questionnaire-See Appendix E)
* Severely reduced life expectancy (e.g., self-reported diagnosis of metastatic cancer, congestive heart failure, or end-stage kidney disease)
* Self-reported diagnosis of sickle cell disease
* Skin damage or rash in the upper arm region where ambulatory blood pressure monitor is to be placed
* Currently enrolled in psychotherapy, and
* Self-reported history or current diagnosis of bipolar disorder, dissociative disorder, psychosis, or substance abuse; or have severe depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Ambulatory Blood Pressure at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  The ambulatory blood pressure monitor (the Spacelabs Healthcare 90217A ABPM) will capture 24-hour daytime and nighttime systolic and diastolic blood pressure reading in the natural environment and will capture heart rate variability. The ambulatory blood pressure monitor will record the subject's systolic and diastolic blood pressure periodically every 30 minutes to one hour and the data will be stored in the internal memory until uploaded to a companion application for visualization and analysis. In addition to ambulatory blood pressure the wearable device will record pulse waves on a beat to beat basis from which heart rate variability will be calculated and analyzed.

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale: Change from Baseline Depressive Symptoms at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  Center for Epidemiological Studies Depression-Scale. The total score is computed. Scores range from 0-60, with higher scores indicating greater symptoms of depression.
Life Orientation Test-Revised: Change from Baseline Dispositional Optimism at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  Life Orientation Test-Revised. Two sub-scale scores are computed for affirming optimism and disaffirming pessimism. Scores range from 0-12 on each sub-scale and summed, with higher scores indicating greater optimism.
General Well-being Schedule: Change in Baseline Emotional Vitality at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  General Well-being Schedule
Life Engagement Test: Change in Baseline Life engagement and Meaning at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  Life Engagement Test
Perceived Stress Scale: Change from Baseline Perceived Stress at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  Perceived Stress Scale. The total score is computed. Scores range from 0 to 16, with higher scores indicating greater perceived stress.
Modified Differential Emotions Scale: Change from Baseline Positive and Negative Affect at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  Modified Differential Emotions Scale. Two sub-scale scores are computed for positive emotions and negative emotions. The sub-scales are averaged, with higher scores indicating higher positive or negative emotions.
Positive Skills: Change in Baseline Positive Skills at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  Positive Skills
Medical Outcomes Study Social Support Survey: Change in Baseline Perceived Social Support at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  Medical Outcomes Study Social Support Survey. Four sub-scale scores are computed for 1) emotional/informational support 2) Tangible support 3) Affectionate Support and 4)Positive Social Interaction. An additional item asks the participant to quantify the number of persons of support. Sub-scale scores range from 1-5, and they are summed for a total score for perceived social support ranging from 0-25, with higher scores indicating greater perceived support.
Medication Adherence: Change in Baseline Medication Adherence at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  Medication Adherence
12-Item Short Form Survey: Change in Self-Reported Mental and Physical Health at 5- and 12-weeks | Baseline, 5-, and 12-weeks
  12-Item Short Form Survey. The total score is computed. Scores range from 0-100, with higher scores indicating greater perceived physical and mental health.

OTHER OUTCOMES:
Physical Activity: Change in Hypertension-related Health Behavior(s) | Baseline, 5-, and 12-weeks
  Self-Reported Physical Activity
Diet: Change in Hypertension-related Health Behavior(s) | Baseline, 5-, and 12-weeks
  Sodium Intake Diet using Scored Sodium Questionnaire. The total score is computed. Scores range from 0-215, with higher scores indicating greater sodium intake.
Change in Heart Rate Variability | Baseline, 5-, and 12-weeks
  Beat-to-beat interval
Change in High-sensitivity C-Reactive Protein | Baseline, 5-, and 12-weeks
  mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Rosalba Hernandez, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- UI Health Pilsen Family Health Center Lower West, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigator will make the data available to users only under a data-sharing agreement that provides for: (1) a commitment to use data only for research purposes and not to identify any individual participant; (2) a commitment to secure the data using appropriate technology; and (3) a commitment to destroy or return data after analyses are completed. If additional outputs result from this research that would be appropriate to share with a wider audience, the investigator will work with the Research Data Service at the University Library to determine appropriate venues for archiving and sharing.
Supporting Information: Study Protocol, ICF
Time Frame: Data may be available by 2022 for a 5-year period.
Access Criteria: The investigator will make the data available to users only under a data-sharing agreement that provides for: (1) a commitment to use data only for research purposes and not to identify any individual participant; (2) a commitment to secure the data using appropriate technology; and (3) a commitment to destroy or return data after analyses are completed. If additional outputs result from this research that would be appropriate to share with a wider audience, the investigator will work with the Research Data Service at the University Library to determine appropriate venues for archiving and sharing.

REFERENCES:
- [Derived] Hernandez R, Cohn M, Hernandez A, Daviglus M, Martinez L, Martinez A, Martinez I, Durazo-Arvizu R, Moskowitz J. A Web-Based Positive Psychological Intervention to Improve Blood Pressure Control in Spanish-Speaking Hispanic/Latino Adults With Uncontrolled Hypertension: Protocol and Design for the inverted exclamation markAlegrate! Randomized Controlled Trial. JMIR Res Protoc. 2020 Aug 4;9(8):e17721. doi: 10.2196/17721. PMID 32749224